CLINICAL TRIAL: NCT03253497
Title: To Evaluate the Effect of Chlorhexidine-benzidamine Administration Prior to the Use of the Laryngeal Mask
Brief Title: To Evaluate the Effect of Chlorhexidine-benzidamine Administration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Savas Altinsoy, Diskapi Yildirim Beyazit Education and Research Hospital anestehesia and reanimation, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: savaş
Record Dates: First submitted 2017-08-11; First posted 2017-08-18 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Effects of Topical Chlorhexidine and Benzidine Spray
Keywords: chlorhexidine, benzidamine, laryngeal mask

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine- benzidamine (Active Comparator): before 15 minute anesthesia induction Chlorhexidine-benzidamine spray will be administrated to oropharynx
  Interventions: Drug: Chlorobenzene Liquid
- Control (No Intervention): before 15 minute normal salin will be administrated to oropharynx

INTERVENTIONS:
Drug: Chlorobenzene Liquid — before induction will be used for oropharynx
  Arms: Chlorhexidine- benzidamine

SUMMARY:
The use of laryngeal mask (LMA) for the purpose of providing airway safety of patients is a common method in general anesthesia practice. This practice does not require laryngoscopy and there is no laryngeal and tracheal stimulation until endotracheal intubation, so an increased hemodynamic response is not expected in the patient. LMA is an airway control device consisting of a silicon mask commonly used in cases where endotracheal intubation (ETE) is not required and a silicone tubing connected by 30 degrees. The glottic settles around the entrance. There is no obligation for muscle relaxation as LMA is intubated. However, if a muscle relaxant agent is not used, pharyngolaryngeal side effects such as patient wounds, hiccups, coughs, involuntary muscle movement, hypoxia, laryngospasm can be seen when LMA is inserted. In these patients complications such as throat burning, sore throat, ear pain, voice anxiety, swallowing difficulties are seen depending on the difficulty of LMA placement in the postoperative period.

Benzidamine is an anti-inflammatory analgesic agent that is not related to the steroid group as the structure. Benzidamine is different from other non-steroidal anti-inflammatory agents in terms of base formation. Benzidamine has local anesthetic effect in concentrations used in topical treatment. Chlorhexidine grams (+) gram (-) bacteria are most effective in microorganisms such as yeast and some fungi and viruses. Chlorhexidine delays bacterial spread with delayed surface effect. It is absorptive from the microbial cell walls and causes membrane leakage.

In this study, investigators aimed to reveal the effects of topical chlorhexidine and benzidamine containing spray (chlorobenzene 30 Ml Spray) used before LMA placement on hemodynamic response with postoperative throat and ear pain, swallowing difficulty, voice anxiety and soft LMA removal.

DETAILED DESCRIPTION:
50 participants with American Society of Anesthesiologists (ASA) physical score I-II. laryngeal mask (LMA) will use in general anesthesia.

all participants will be premedicated with 0.05 mg/kg midazolam 30 minutes before the operation. ASA, age, sex, body mass index (BMI) will record. peripheral oxygen saturation (SaO2) ,electrocardiography and non invasive blood pressure will monitored. A venous cannula will place on the back of the hand. participants will randomly divide into 2 groups by closed envelope method.

before 15 minute anesthesia induction topical chlorobenzene 30 Ml Spray will use. Than LMA will placement on and record hemodynamic response and postoperative throat and ear pain, swallowing difficulty, voice anxiety and soft LMA removal.

ELIGIBILITY:
Inclusion Criteria:

* general anesthesia

Exclusion Criteria:

* using anti-inflammatory drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-09-02 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2017-12-02 (Actual)

PRIMARY OUTCOMES:
Removal to soft LMA | First minute after extubation
  was assessed because of coughing, tooth clenching, desaturation, and lack of laryngeal spasm
complications | after operation 1th, 6th, 12th and 24th hour
  sore throat, ear pain, swallowing difficulty, nausea and vomiting

SECONDARY OUTCOMES:
hemodynamic response | before LMA and at 1 minute after LMA applied
  systolic, diastolic and mean blood pressure will record before LMA and post LMA used at first minute.
Heart rate | before LMA and at 1 minute after LMA applied
  Heart rate will record before LMA insertion and post LMA used at first minute.

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health Diskapi Yıldırım Beyazıt Training and Research Hospital, Ankara, Turkey (Türkiye)